CLINICAL TRIAL: NCT05073692
Title: Comparison of Type 2 Diabetes Pharmacotherapy Regimens Using Targeted Learning
Brief Title: Comparison of Type 2 Diabetes Pharmacotherapy Regimens
Acronym: ON TARGET DM
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Geisinger Clinic (Other); Henry Ford Health System (Other); HealthPartners Institute (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 739857
Record Dates: First submitted 2021-09-14; First posted 2021-10-11 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Diseases
Keywords: Type 2 Diabetes Mellitus; Cardiovascular Diseases; Medication; Treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Linagliptin; Exenatide; Liraglutide; empagliflozin; glimepiride; Glipizide; alogliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: SU — Exposure to the class of drugs known as Sulfonylureas (SU)
Drug: DPP4 — Exposure to the class of drugs known as Dipeptidyl peptidase-4 inhibitors (DPP4)
Drug: SGLT2i — Exposure to the class of drugs known as Sodium-glucose cotransporter-2 inhibitors (SGLT2i)
Drug: GLP-1RA — Exposure to the class of drugs known as Glucagon-like peptide-1 receptor agonists (GLP-1RA)
Drug: SGLT2i or GLP-1RA — Exposure to either SGLT2i or GLP-1RA
Drug: Linagliptin (DPP4) — Exposure to agent Linagliptin (DPP4)
Drug: Exenatide (GLP-1RA) — Exposure to agent Exenatide (GLP1-RA)
Drug: Liraglutide (GLP-1RA) — Exposure to agent Liraglutide (GLP-1RA)
Drug: Empagliflozin (SGLT2i) — Exposure to agent Empagliflozin (SGLT2i)
Drug: Glimepiride (SU) — Exposure to agent Glimepiride (SU)
Drug: Glipizide (SU) — Exposure to Glimepiride (SU)
Drug: Glimepiride (SU) or Glipizide (SU) — Exposure to agent Glimepiride (SU) or Glipizide (SU)
Drug: SU or DPP4 (excluding saxagliptin and alogliptin) — Exposure to either SU or DPP4 excluding Saxagliptin and Alogliptin
Drug: Exenatide (GLP-1RA) or Liraglutide (GLP-1RA) — Exposure to either Exenatide (GLP-1RA) or Liraglutide (GLP-1RA)

SUMMARY:
This study is designed to help patients with type 2 diabetes and their clinicians: (a) identify which glucose lowering medications have the most favorable effects on heart health and other patient-important outcomes, (b) inform the timing of medication initiation, and (c) identify whether medication benefits apply equally to all adults with type 2 diabetes, or may be different based on age, sex, race/ethnicity, baseline heart health status, baseline renal function, or other factors.

DETAILED DESCRIPTION:
The study will conduct head-to-head comparisons of type 2 diabetes mellitus (T2DM) treatment strategies using observational data from real-world clinical settings to assess cardiovascular disease (CVD) outcomes and other patient-centered outcomes in T2DM patients with moderate baseline CVD risk who are treated with each of these four classes of glucose-lowering medications known as SGLT2, GLP-1RA, DPP4, and SU. To mitigate bias concerns related to confounding and informative loss to follow-up, analyses will be based on modern causal inference methods combined with machine learning that emulate intention-to-treat (ITT) and per-protocol (PP) analyses of pragmatic randomized trials with active comparators to provide the most robust and precise estimates of relative and absolute effects we would expect in usual care settings.

Specific Aims and Hypotheses:

Aim 1. Compare the effect off SGLT21, GLP-1RA, DPP4, and SU on each study outcome in adults with T2DM when each type of medication is (a) initiated as second-line therapy after metformin, and (b) initiated as first-, second-, or third-line therapy, or after any history of glucose-lowering therapy independent of prior metformin use.

Aim 2. Compare the effect on each study outcome of earlier versus later initiation of SGLT2i, GLP-1RA, DPP4, SU as first-, or second-, or third-line therapy, or after any history of glucose-lowering therapy triggered by various changes in A1C, or CVD risk, or other patient characteristics.

Aim 3. Assess in each of the prior analyses whether the treatment effects on study outcomes vary across categories of baseline CVD risk and CVD event history, renal function, congestive heart failure status, age, sex and race/ethnicity, or other patient characteristics.

Glucose-lowering medications will be compared at both the class and agent level. The key outcomes that will be considered are MACE 3-point, Myocardial Infarction, Stroke, Heart Failure, Hospitalization, Coronary or Carotid Artery Stent or Bypass Procedure, CVD Mortality, Overall Mortality. Additional patient-centered outcomes will be specified based on insights from stakeholder members of the research team.

ELIGIBILITY:
* Dispensing of either of the set of drugs being compared
* No prior dispensing of nor contraindication for any of the drugs compared
* Evidence of Type 2 Diabetes Mellitus diagnosis
* Age 18 or older
* Not currently pregnant
* No evidence of dementia or short-term life expectancy from prior cancer diagnoses
* History of ≥2 years of continuous health plan membership
* ≥1 A1c test in the past 18 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from six large care delivery systems with integrated administrative and EHR clinical data sources (Geisinger in Pennsylvania, Henry Ford Health System in Michigan, HealthPartners Institute in Minnesota and Wisconsin, and Kaiser Permanente of Northern California, Southern California, and Hawaii) who were new users of glucose-lowering medications between 01/01/2014 and 12/31/2021.
Sampling Method: Non-Probability Sample
Enrollment: 241981 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Romain S. Neugebauer, PhD, Principal Investigator — Kaiser Permanente; Patrick J O'Connor, MD, MA, MPH, Principal Investigator — HealthPartners Institute
Locations (6):
- United States (6):
  - Kaiser Permanente Southern California, Pasadena, California
  - Romain S. Neugebauer, Pleasanton, California
  - Kaiser Permanente Hawaii, Honolulu, Hawaii
  - Henry Ford Health System, Detroit, Michigan
  - HealthPartners Institute, Bloomington, Minnesota
  - Geisinger, Danville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomas TW, Hooker SA, Schmittdiel JA. Principles for Stakeholder Engagement in Observational Health Research. JAMA Health Forum. 2024 Mar 1;5(3):e240114. doi: 10.1001/jamahealthforum.2024.0114. PMID 38488777
- [Result] Rodriguez LA, Finertie H, Neugebauer RS, Gosiker B, Thomas TW, Karter AJ, Gilliam LK, Oshiro C, An J, Simonson G, Cassidy-Bushrow AE, Dombrowski S, Nolan M, O'Connor PJ, Schmittdiel JA. Race and ethnicity and pharmacy dispensing of SGLT2 inhibitors and GLP-1 receptor agonists in type 2 diabetes. Lancet Reg Health Am. 2024 May 7;34:100759. doi: 10.1016/j.lana.2024.100759. eCollection 2024 Jun. PMID 38745886
- [Result] Thapa B, Schmittdiel JA, Arterburn D, Neugebauer R, Dyer W, O'Connor PJ, An J, Cassidy-Bushrow AE, Gilliam LK, Hooker SA, Nolan MB, Oshiro CES, Thomas T, Simonson G, Dombrowski SK, Rodriguez LA. Clinical and Demographic Characteristics Associated With Diabetes Remission in Six Integrated Health Care Systems: A Retrospective Cohort Study. Diabetes Care. 2025 Oct 1;48(10):1737-1743. doi: 10.2337/dc25-0530. PMID 40734551
- [Result] Neugebauer R, An J, Dombrowski SK, Oshiro C, Cassidy-Bushrow A, Gilliam L, Simonson G, Karter AJ, Bergenstal R, Finertie H, Yassin MM, Knowlton G, Lin SR, Dyer W, Pimentel N, Izadian K, Schmittdiel J, Thomas TW, Hooker SA, Nolan MB, Wright E, Aurora L, Rodriguez LA, Kaur J, Adams AS, van der Laan MJ, O'Connor PJ. Glucose-Lowering Medication Classes and Cardiovascular Outcomes in Patients With Type 2 Diabetes. JAMA Netw Open. 2025 Oct 1;8(10):e2536100. doi: 10.1001/jamanetworkopen.2025.36100. PMID 41091469

RESULTS

PARTICIPANT FLOW:
Groups:
- SU Initiators: Initiators of Sulfonylurea between 01/01/2014 and 12/31/2021; sample size N=212,042.
- DPP4 Initiators: Initiators of DPP4 between 01/01/2014 and 12/31/2021; sample size N=5,862.
- SGLT2i Initiators: Initiators of SGLT2i between 01/01/2014 and 12/31/2021; sample size N=14,858.
- GLP-1RA Initiators: Initiators of GLP-1RA between 01/01/2014 and 12/31/2021; sample size N=9,219.
Period: Overall Study
Arm/Group | SU Initiators | DPP4 Initiators | SGLT2i Initiators | GLP-1RA Initiators
Started | 212042 | 5862 | 14858 | 9219
Completed | 169348 | 4402 | 13681 | 7863
Not Completed | 42694 | 1460 | 1177 | 1356

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SU Initiators | DPP4 Initiators | SGLT2i Initiators | GLP-1RA Initiators | Total
Number analyzed (Participants) | 212,042 | 5,862 | 14,858 | 9,219 | 241981
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.91 (12.91) | 61.69 (12.88) | 60.51 (11.95) | 55.95 (12.34) | 57.21 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95,560 | 3,123 | 6,537 | 5,319 | 110539
  Male | 116,482 | 2,739 | 8,321 | 3,900 | 131442
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 78,965 | 1,098 | 3,501 | 1,943 | 85507
  Not Hispanic or Latino | 133,077 | 4,764 | 11,357 | 7,276 | 156474
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1,505 | 26 | 92 | 48 | 1671
  Asian | 33,756 | 735 | 2,690 | 731 | 37912
  Native Hawaiian or Other Pacific Islander | 3,303 | 61 | 371 | 143 | 3878
  Black or African American | 20,977 | 669 | 1,483 | 1,343 | 24472
  White | 103,428 | 3,689 | 7,666 | 5,609 | 120392
  More than one race | 5,740 | 186 | 662 | 523 | 7111
  Unknown or Not Reported | 43,333 | 496 | 1,894 | 822 | 46545

OUTCOME MEASURES:

1. Primary Outcome: Incidence of 3-point Major Adverse Cardiovascular Events (MACE)
Description: 3-point MACE is defined as a single outcome measure, which is a composite measure of nonfatal myocardial infarction, nonfatal stroke, or cardiovascular disease death.
Time Frame: 2.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | SU Initiators | DPP4 Initiators | SGLT2i Initiators | GLP-1RA Initiators
Number analyzed (Participants) | 212,042 | 5,862 | 14,858 | 9,219
Participants | 11,348 | 393 | 424 | 296

ADVERSE EVENTS:
Time Frame: 2.5 years.
Description: Death other than cardiovascular death which is included in the study primary outcome MACE. We are reporting these deaths as all-cause mortality.
  No Other Adverse Events or Serious Adverse Events were defined as part of this observational study and its protocol.
  Serious and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | SU Initiators | DPP4 Initiators | SGLT2i Initiators | GLP-1RA Initiators
All-Cause Mortality (participants affected / at risk) | 4867/212042 | 235/5862 | 117/14858 | 109/9219
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT05073692/Prot_SAP_000.pdf